CLINICAL TRIAL: NCT01582113
Title: Cognizin Citicoline Dosing in a Healthy Adolescent Male Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Deborah Yurgelun-Todd (Other)
Responsible Party: Sponsor-Investigator, Deborah Yurgelun-Todd, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_49504
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Neurocognitive Improvement
MeSH Terms: interventions — Cytidine Diphosphate Choline; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Citicoline (Experimental): At visit 1 and again at visit 2, participants assigned to the experimental arm will receive a 14-day supply of 500 mg of citicoline, of which they will be instructed to take 500 mg daily. This will be done in a double-blind, randomized fashion.
  Interventions: Drug: Citicoline
- Low Dose Citicoline (Experimental): At visit 1 and again at visit 2, participants assigned to the experimental arm will receive a 14-day supply of 250 mg of citicoline, of which they will be instructed to take 250 mg daily. This will be done in a double-blind, randomized fashion.
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): At visit 1 and again at visit 2, participants assigned to the placebo group will be given 14-day supplies of placebo to be taken daily throughout the study period. This will be done in a double-blind, randomized fashion.
  Interventions: Other: Microcrystalline Cellulose

INTERVENTIONS:
Drug: Citicoline — Participants randomly assigned to the experimental group, who, in addition to the research staff will be blind to such assignment, will be instructed to orally administer 500 mg or 250 mg daily citicoline. These participants will receive a 14-day supply of citicoline at visit 1 and again at visit 2, making for a 28-day administration period.
  Other Names: Cognizin Citicoline
  Arms: High Dose Citicoline; Low Dose Citicoline
Other: Microcrystalline Cellulose — Microcrystalline Cellulose will be the placebo administered to participants randomly assigned to the placebo arm. Microcrystalline Cellulose will serve as the placebo for Citicoline and will be orally administered daily in 470 mg doses.
  Arms: Placebo

SUMMARY:
To determine the functional effects of Citicoline, a natural supplement, when administered for a duration of four weeks (28 days) to non-psychiatric adolescent male participants. The investigators hypothesize that citicoline will provide cognitive benefits to this population after 28 days of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 13-18 years old
* No history of co-morbid psychiatric disorder, current Axis I or II diagnosis or previous pharmacotherapeutic trial

Exclusion Criteria:

* Head injury with LOC > 5 minutes
* Use of any psychotropic medication

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2012-06; Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Neurocognitive performance | 28 days
  Using baseline assessment measures gathered at Visit 1, assessments collected at Visits 2 and 3 will be used to determine whether the combined administration of citicoline will improve neurocognitive performance in male adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- The Brain Institute, University of Utah, Salt Lake City, Utah, United States